CLINICAL TRIAL: NCT04336930
Title: Evaluation of the Pupillary Dilatation Reflex With the "Pupillary Pain Index" in Neurological Prognosis After Cardiac Arrest
Brief Title: Evaluation of the "Pupillary Pain Index" in Neurological Prognosis After Cardiac Arrest
Acronym: CAPPI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI275
Record Dates: First submitted 2020-03-10; First posted 2020-04-07 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Arrest; Post-Anoxic Coma; Anoxic Brain Injury
Keywords: Pupillometry; Pupillary Pain Index; Brain ischemia; Heart arrest; Neuroprognostication
MeSH Terms: conditions — Heart Arrest; Hypoxia-Ischemia, Brain; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Arrest group: Patients remaining comatose after a cardiac arrest
  Interventions: Diagnostic Test: Pupillary pain index (PPI)

INTERVENTIONS:
Diagnostic Test: Pupillary pain index (PPI) — Measurement of PPI with a pupillometer

SUMMARY:
Two-thirds of patients admitted to the Intensive Care Unit after a cardiac arrest die in the context of treatment withdrawal after a multimodal evaluation that determines an unfavorable neurological outcome.

This study will evaluate the Pupillary Pain Index (PPI) in the neurological prognosis after cardiac arrest. The PPI is determined by recording of pupillary dilatation with a videopupillometer after a calibrated and incremented nociceptive stimulus on a cutaneous metamere.

DETAILED DESCRIPTION:
Cardiorespiratory arrest is associated with high mortality and morbidity rates. The direct consequence of a cardio-circulatory arrest is the absence of blood flow allowing oxygenation of the organs and consequently formation of ischemic lesions. Anoxic cerebral lesions are common in the aftermath of a cardiac arrest and often lead to the death of patients when active therapies are stopped after a multimodal prognostication that indicates that a poor outcome is very likely.

It is of paramount importance to optimize the sensitivity of the prognostication strategy in detecting good neurological outcome. A multimodal approach to the prognostic assessment is essential, and must include at least clinical examination, electrophysiology exploration (electroencephalography and/or evoked potentials) and biomarker analysis.

Although the most reliable predictors did not give false positives in most studies, none of them, considered individually, can establish an unfavorable prognosis with an absolute degree of certitude. For these reasons it is interesting to evaluate new prognostication tools.

The videopupillometry allows precise, reproducible and repeated measurement of changes in pupil diameter in response to a painful or a luminous stimulus. Pupillary pain reflex analysis is usually used to assess the degree of analgesia in a non-communicative patient during general anesthesia and neuromuscular blockade. The PPI score is determined at the bedside by recording pupillary dilatation after a calibrated and incremented nociceptive stimulus (electrical current between 5 and 60mA) applied to a skin metamere with two electrodes.

Automated pupillometry measurement has been recently developed to help support prognostication, with a quantitative pupillary light reflex measurement. The aim of this study is to evaluate the Pupillary Pain Index in the neurological prognosis after a cardiac arrest by correlating the PPI at 48h from the patient's arrival to the CPC score at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU after cardiac arrest
* Age > 18 years
* Presenting a Glasgow score of <8 at admission

Exclusion Criteria:

* Pregnancy
* Ocular pathology making pupillometry impossible.
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients remaining comatose after cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Score Cerebral Performance Category (CPC) | 3 months
  Good outcome defined as CPC 1-2, poor outcome defined as CPC 3-5

SECONDARY OUTCOMES:
Characteristics of electroencephalography pattern | Day 2, day 3, day 5, day 7
  Classification of Synek, type of pattern (Very malignant, malignant or benign)
Biomarkers | 24 hours, 48 hours
  Value of seric Neuron Specific Enolase
Glasgow motor score | 24 hours, 48 hours, day 5, day 7
  Motor response component of the Glasgow Coma Scale, ranging from 1 (no response) to 6 (normal response)
ICU parameters | Day 14
  Ventilator days, Length of stay
Evoked Potentials | Day 14
  Presence or absence of the N20 component of the evoked potentials
Neurological pupil index | Day 2, day 3
  standardized evaluation of pupil reactivity ranging from 0 (sluggish or abnormal pupils) to 5 (normally reactive pupils)
Diameter of the pupil | 24 hours, 48 hours, 72 hours
  In millimeters (pupillometry measure)
Percentage of pupil dilatation | 24 hours, 48 hours, 72 hours
  Pupillometry measure
Latency of pupil dilatation | 24 hours, 48 hours, 72 hours
  In milliseconds (pupillometry measure)
Velocity of pupil dilatation | 24 hours, 48 hours, 72 hours
  In millimeters per second (pupillometry measure)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Koszutski, Dr, Principal Investigator — Nancy Teaching Hospital, CHU de Nancy

IPD SHARING:
Plan to Share IPD: No